CLINICAL TRIAL: NCT05197257
Title: 68Ga-PSMA-11 PET in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-4070.cc
Record Dates: First submitted 2021-12-16; First posted 2022-01-19 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Newly Diagnosed
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Men with pathologically proven prostate adenocarcinoma (Experimental): The intervention is a PET scan with the radiolabelled PSMA ligand, 68Ga-PSMA-11. The PET may be combined with a CT scan as a PET/CT or an MRI scan as PET/MRI. 68Ga-PSMA-11 PET/CT will be acquired using a modern digital GE PET/CT scanner or a modern digital PET / MRI scanner.
  Interventions: Drug: Ga-PSMA-11

INTERVENTIONS:
Drug: Ga-PSMA-11 — The PSMA Sterile Cold Kit, is a kit comprising all needed materials (lyophilized PSMA for PSMA reconstitution, elution vial for Ga and ancillary materials for transfer between vials) to perform a room-temperature radiolabelling of PSMA-11 with Ga. Ga is not part of the kit and should be provided in the form gallium chloride solution following the requirements of the relevant local regulations. PSMA-11 radiolabelled with Ga is administered in patients with prostate cancer recurrence after radical treatment.

SUMMARY:
Patients will receive a single dose of 68Ga-PSMA-11 and undergo a PET/CT or PET/MRI imaging study.

DETAILED DESCRIPTION:
This is a prospective, Phase III, single-center, open-label to provide extended access in patients with biochemically recurrent prostate cancer. Approximately 100 patients are planned for enrollment in this study. Patients will receive a single dose of 68Ga-PSMA-11 and undergo a PET/CT or PET/MRI imaging study.

The intervention is a PET scan with the radiolabelled Prostate-specific membrane antifen (PSMA) ligand, 68Ga-PSMA-11. The PET may be combined with a CT scan as a PET/CT or an MRI scan as PET/MRI. 68Ga-PSMA-11 PET/CT will be acquired using a modern digital GE PET/CT scanner or a modern digital PET / MRI scanner.

AEs will be collected during injection and uptake phase (45-120 min posts infusion) of Ga-68 PSMA-11 PET/CT scan. All safety events will be recorded up to 120 min post injection.

Men with pathologically proven prostate adenocarcinoma, high risk cancer at diagnosis, evidence of biochemical recurrence, or known metastatic disease planned to start and change systemic therapy regimen.

One intravenous catheter will be placed for radiopharmaceutical administration. Patients will be injected with 100 MBq (3mCi)-300 MBq( 7mCi) of 68Ga-PSMA-11 via this catheter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven prostate adenocarcinoma
* Age ≥ 18 years
* Patients already diagnosed with prostate cancer: Primary Staging: intermediate and high-risk patients per NCCN guidelines
* Biochemical Recurrence: Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy):

  a. Post radical prostatectomy (RP) - AUA recommendation i. PSA greater than or equal to 0.2 ng/mL measured more than 6-13 weeks after RP and confirmed by a second determination of a PSA level of >0.2 ng/mL b. Post-radiation therapy - ASTRO-Phoenix consensus definition i. Nadir + greater than or equal to 2 ng/mL rise in PSA
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Unable to lie flat, still or tolerate a PET/CT scan, or any other condition that would preclude PET/CT imaging.
* Patients with any medical condition or circumstance that the investigator believes may compromise the data collection or lead to a failure to fulfil the study requirements.
* Patients with known hypersensitivity to the active substance or to any of the excipients of the investigational product.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 39 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett Chin, Principal Investigator — Colorado Research Center
Locations (2):
- United States (2):
  - Colorado Research Center, Aurora, Colorado
  - UCHealth-Metro Denver, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Men With Pathologically Proven Prostate Adenocarcinoma
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Men With Pathologically Proven Prostate Adenocarcinoma
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse Events (AEs) will be collected and reviewed to monitor for safety. Incidence and severity of AEs and adverse events will be estimated with 95% confidence intervals summarized with descriptive statistics. CTCAE version 5.0 will be used to grade AEs.
Time Frame: Immediately after administration and for 1 hour and 30 minutes afterwards
Population: All patients observed for safety.
Measure: Count of Participants; unit: Participants
Groups:
- Adverse Events- All Grades: Number of Adverse Events (all grades) observed immediately after administration and for 1 hour and 30 minutes afterward.
Arm/Group | Adverse Events- All Grades
Number analyzed (Participants) | 39
Participants | 0

2. Secondary Outcome: Compare the Diagnostic Impact of 68Ga-PSMA-11 PET/CT Imaging Over Current Standard of Care Imaging Modalities.
Description: Determine the frequency of positive PSMA PET scans in relation to the PSA value before the PSMA scans and compared to conventional imaging. Results will be summarized descriptively with 95% confidence intervals. Determine rate of overall changes in management by comparing planned management strategy using conventional imaging with executed management strategy incorporating information from 68Ga-PSMA-11 PET/CT, regardless of treatment modality.
  Analysis: The rate of change in management based on the incorporation of68Ga-PSMA-11 PET/CT results will be expressed as the percentage of total patients imaged in which change in management occurred, regardless of treatment modality. The rate of change in management will also be estimated within each group (initial staging, biochemical recurrence, and pre/post treatment). 95% confidence intervals (CIs) will be used to express precision of the estimates.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Groups:
- Initial Treatment Strategy Group With PSMA Uptake: Patients with newly diagnosed with prostate cancer: Primary Staging: high / intermediate risk per NCCN guidelines.
  Count of patients with newly diagnosed prostate cancer who showed PSMA uptake in either in the prostate or in metastatic lesions.
- Initial Treatment Strategy Group- Patient Management: Count of participants with newly diagnosed with prostate cancer whose providers changed the clinical management plan after review of the PSMA PET/CT results.
- Subsequent Treatment Strategy Group: Biochemical Recurrence: Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy) or other local therapies.
  Count of participants whose PSMA PET showed more prostate cancer lesions compared to conventional imaging.
- Subsequent Treatment Strategy Group- Patient Management: Count of participants whose PSMA PET/CT scans significantly changed patient management plan
- All Participants- Initial and Subsequent Strategy: Count of all study participants whose PSMA PET/CT scans did not show additional lesions compared to conventional imaging.
Arm/Group | Initial Treatment Strategy Group With PSMA Uptake | Initial Treatment Strategy Group- Patient Management | Subsequent Treatment Strategy Group | Subsequent Treatment Strategy Group- Patient Management | All Participants- Initial and Subsequent Strategy
Number analyzed (Participants) | 12 | 12 | 27 | 27 | 39
Participants | 12 | 1 | 22 | 21 | 7

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | Men With Pathologically Proven Prostate Adenocarcinoma
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT05197257/Prot_SAP_ICF_000.pdf